A Randomised, Cross-Over, Single-Blind, Relative Bioavailability Study of Nicotine Delivery From Selected Oral Nicotine Products

NCT05452278

Statistical Analysis Plan Final Version 1.0 – 23 Nov 2021



# CONFIDENTIAL

# Statistical analysis plan (SAP)

| Sponsor: | Imperial Tobacco Ltd |
|---|---|
| Study code: | IB-OND-ZONEX-11 |
| CTC project no: | 369-62-2021 |
| Study title: | A RANDOMISED, CROSS-OVER, SINGLE-BLIND, RELATIVE BIOAVAILABILITY STUDY OF NICOTINE DELIVERY FROM SELECTED ORAL NICOTINE PRODUCTS |
| SAP version and date: | Final version 1.0 23NOV2021 |
| CTC biostatistician: | |

Protocol Version No: Final v1.0; 21JUN2021

Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



## 1 TABLE OF CONTENTS

| 1 | T | ABLE OF CONTENTS | 2 |
|---|---|---|---|
| 2 | V | ERSION HISTORY | 5 |
| 3 | I | NTRODUCTION | 5 |
| 4 | C | CLINICAL STUDY DETAILS | 5 |
| | 4.1 | Clinical study objectives and endpoints | 5 |
| | 4.2 | Clinical study design | 6 |
| | 4.3 | Statistical hypotheses | 7 |
| | 4. | .3.1 Statistical hypotheses related to primary objective | 7 |
| | 4.4 | Number of subjects | 7 |
| | 4.5 | Randomisation | 7 |
| | 4.6 | Blinding | 7 |
| 5 | S | TATISTICAL AND ANALYTICAL PLANS | 8 |
| | 5.1 | Sample size determination | 8 |
| | 5.2 | Definition of analysis sets | 8 |
| | 5. | .2.1 Full analysis set | 8 |
| | 5. | .2.2 Pharmacokinetic analysis set | 8 |
| | 5. | .2.3 Use of analysis set | 8 |
| | 5.3 | Definition of baseline | 8 |
| | 5.4 | Output rounding principles | 8 |
| | 5.5 | Significance level | 9 |
| | 5.6 | Multiple comparisons/multiplicity | 9 |
| | 5.7 | Handling of dropouts, missing data and outliers | 9 |
| 6 | P | HARMACOKINETIC ANALYSIS | 9 |
| 7 | C | CLINLCAL DATABASE PROCESSING | . 11 |
| | 7.1 | General information | . 11 |
| | 7.2 | Database modeling of study design | 11 |
| 8 | S | TATISTICAL METHODOLOGY | . 12 |
| | 8.1 | Primary endpoint(s) analysis | 12 |
| | 8. | .1.1 C <sub>max</sub> and AUC <sub>t</sub> | |
| | 8. | .1.2 Tables and Figures relating to the primary endpoint(s) | 12 |
| | 8.2 | Secondary endpoint(s) analysis | 13 |
| | 8. | .2.1 Definition of endpoint(s) | . 13 |
| | 8. | .2.2 Tables and Figures relating to the secondary endpoint(s) | . 15 |


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



| | 8.3 | Tertiary/exploratory endpoint(s) analysis | 17 |
|---|---|---|---|
| | 8.4 | Other data analysis/presentation | 17 |
| | 8.4 | 4.1 Demographics and baseline characteristics | 17 |
| | 8. | 4.2 Medical/surgical history and prior/concomitant medication | 17 |
| | 8.5 | Interim analysis | . 17 |
| 9 | <b>C</b> ] | HANGES FROM THE CSP | . 17 |
| | 9.1 | Changes of product comparisons for primary analysis | . 17 |
| | 9.2 | Changes of fixed effects for primary analysis | 18 |
| | 9.3 | Change of analysis method for Urge to use questionnaire for secondary analysis | 18 |
| 1 | 0 | STATISTICAL DELIVERABLES | 18 |
| 1 | 1 | SOFTWARE | 18 |
| 1 | 2 | APPROVAL | 19 |
| 1. | 3 | SUPPORTIVE DOCUMENTATION | 20 |
| | 13.1 | Appendix 1 – list of abbreviations | 20 |
| 1 | 4 | STATISTICAL OUTPUT LAYOUT | 21 |
| | 14.1 | Template tables | 21 |
| | Те | emplate table A Descriptive statistic table – continuous variables | 22 |
| | Te | emplate table B Descriptive statistic table – discrete variables | 23 |
| | 14.2 | Template figures | 24 |
| | Те | emplate figure A Subject measurements over time by treatment figure | 24 |
| | Τe | emplate figure B Treatment measurements over time by subject figure | 25 |
| | | emplate figure C Measurements over time by treatment with confidence interval bars gure 26 | 5 |
| | _ | Tables | . 27 |
| | 14.4 | | |
| | 14.5 | | |
| | Li | sting 16.2.1.1. Discontinued subjects (All subjects) | . 46 |
| | Li | sting 16.2.2.1. Protocol deviations (All subjects) | 46 |
| | Li | sting 16.2.3.1 Subjects excluded from PKAS (All subjects) | 46 |
| | Li | sting 16.2.3.2 Population definitions (All subjects) | 46 |
| | Li | sting 16.2.3.3. Non-eligible subjects (All subjects) | . 46 |
| | Li | sting 16.2.4.1. Demography (Full analysis set) | 46 |
| | Li | sting 16.2.4.2 Medical/surgical history (Full analysis set) | 46 |
| | Li | sting 16.2.5.1. Prior and concomitant medications (Full analysis set) | 46 |


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



| Listing 16.2.7.1. HIV, hepatitis B and C (All subjects) | 46 |
|---|---|
| Listing 16.2.8.1. Other laboratory measurements (All subjects) | 46 |
| Listing 16.2.9.2. Product evaluation scale (PES) (Full analysis set) | 46 |
| Listing 16.2.9.3. Urge to use questionnaire (Full analysis set) | 47 |
| Listing 16.2.9.4. Products preference scale (PPS) (Full analysis set) | 47 |
| Listing 16.2.10.1. Plasma concentration (Pharmacokinetic analysis set) | 47 |
| Listing 16.2.10.2. PK parameters (Pharmacokinetic analysis set) | 47 |
| Listing 16.2.19.1. Nicotine pouch collection (Pharmacokinetic analysis set) | 47 |
| Listing 16.2.12.1. Adverse events, part 1 (Full analysis set) | 47 |
| Listing 16.2.12.2. Adverse events, part 2 (Full analysis set) | 47 |
| Listing 16.2.12.3. Serious adverse events, part 1 (Full analysis set) | 47 |
| Listing 16.2.12.3. Serious adverse events, part 2 (Full analysis set) | 47 |
| Listing 16.2.12.4. Serious adverse events, seriousness criteria (Full analysis set) | 47 |
| Listing 16.2.13.1. Safety laboratory (Full analysis set) | 47 |
| Listing 16.2.14.1. Vital signs (Full analysis set) | 47 |
| Listing 16.2.15.1. ECG (Full analysis set) | 47 |
| Listing 16.2.16.1. Physical examinations (Full analysis set) | 48 |
| Listing 16.2.17.1. Disposition (All subjects) | 48 |
| Listing 16.2.18.1. Subject visits (All subjects) | 48 |
| Listing 16.2.19.1. Subject elements (All subjects) | 48 |


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



### 2 VERSION HISTORY

This statistical analysis plan (SAP) for study IB-OND-ZONEX-11 is based on the protocol dated 21JUN2021.

Table 1 SAP version history summary

| SAP version | Approval<br>Date | Changes | Rationale |
|-------------|------------------|---------|-----------------------------------|
| 0.1 | 08NOV2021 | - | Version ready for internal review |
| 0.2 | 10NOV2021 | | Version ready for Sponsor review |
| 1 | 23NOV2021 | NA | Original version |

### 3 INTRODUCTION

This SAP gives details regarding the statistical analyses and data presentation outlined in the final clinical study protocol (CSP) for the study IB-OND-ZONEX-11. Any changes from the final CSP are given in Section 9.

### 4 CLINICAL STUDY DETAILS

## 4.1 Clinical study objectives and endpoints

Table 2 Clinical study objectives and endpoints

| Objectives | Estimands/Endpoints |
|---|---|
| Primary | |
| To evaluate and compare the maximum plasma concentration (C <sub>max</sub> ) and the area under the curve at the last timepoint measured (AUC <sub>t</sub> ) of nicotine after the use of each product. | 1.1 C <sub>max</sub> and AUC <sub>t</sub> |
| Secondary | |
| 2.1 To evaluate other PK parameters of nicotine after the use of each product. | 2.1.1 AUC timepoint 0 to 90 minutes (AUC <sub>0-90</sub> ), AUC timepoint 0 to infinity (AUC <sub>inf</sub> ), time to C <sub>max</sub> (T <sub>max</sub> ), plasma concentration at last timepoint measured (C <sub>last</sub> ), and terminal elimination half-life (T <sub>1/2</sub> ). |
| 2.2 To evaluate orally extracted dose of nicotine in used products (oral nicotine delivery [OND]). | 2.2.1 The orally extracted dose of nicotine from each pouch will be calculated to evaluate the correlation between baseline- |


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



| | adjusted AUC <sub>inf</sub> and orally extracted dose of nicotine. |
|---|---|
| 2.3 To evaluate product perception and preference by use of subjective assessments. | 2.3.1 Subjective assessment endpoints including: Product evaluation scale (PES), Product preference scale (PPS) and the Urge to use questionnaire. |
| 2.4 To evaluate the tolerability and safety of each of the products used. | <ul> <li>2.4.1 Frequency, intensity and seriousness of adverse events (AEs).</li> <li>2.4.2 Clinically significant changes in laboratory parameters, vital signs and electrocardiogram (ECG).</li> </ul> |
| Tertiary/Exploratory | |
| NA | NA |

### 4.2 Clinical study design

This will be a randomised, cross-over, single-blind, confinement study conducted in 27 male or female snus or nicotine pouch users. The study will investigate 4 different nicotine containing products in a cross-over design, incorporating pharmacokinetic (PK) evaluation, nicotine extraction evaluation, subjective questionnaire assessments as well as safety and tolerability evaluation.

During the study participation, subjects will come for 2 visits to the clinic, including a screening visit and a 4-day confinement period. A final follow up end-of-study telephone call will be performed within a week of last product use.

The following figure gives an overview of the study design:




Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



### 4.3 Statistical hypotheses

#### 4.3.1 Statistical hypotheses related to primary objective

The main statistical hypothesis that will be tested in the study is that  $AUC_t$  and  $C_{max}$  does not significantly differ for test product A-B respectively in comparison to product D (Le., the primary objective will be examined by the following statistical comparisons for  $AUC_t$  and  $C_{max}$ :

- Product A does not significantly differ from Product D
- Product B does not significantly differ from Product D
- Product C does not significantly differ from Product D

More information about the statistical tests to be performed can be found in Section 8.1.

### 4.4 Number of subjects

Approximately 54 subjects will be screened to achieve a total of 27 randomised subjects.

#### 4.5 Randomisation

On Day 1, subjects will be randomised to one of 4 treatment sequences. The 4 different products are:

| • A: ZoneX | nicotine/pouch |
|------------|--------------------------------------|
| • B: ZoneX | nicotine/pouch |
| • C: ZoneX | nicotine/pouch |
| • D: | nicotine/ pouch (comparator product) |

The 4 randomisation sequences are described in the table below:

| Sequence | | Oro | der | |
|------------|---|-----|-----|---|
| Sequence 1 | A | В | С | D |
| Sequence 2 | В | C | D | A |
| Sequence 3 | С | D | A | В |
| Sequence 4 | D | A | В | C |

A computer-generated randomisation list will be created by CTC using SAS Proc Plan, SAS Version 9.4 (or later). The randomisation list will contain subject number, sequence and treatment and will be kept by the randomiser until database lock. A copy of the randomization list will be provided to the research clinic.

### 4.6 Blinding

This is a single-blind study, i.e., the Investigator and study staff, but not the subjects, will know the identity of each IP.


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



The IP:s differ somewhat in size but are otherwise identical in appearance. The subjects will not know the strength/nicotine content of each IP.

#### 5 STATISTICAL AND ANALYTICAL PLANS

### 5.1 Sample size determination

No formal sample size calculation has been performed for this study. The proposed sample size is considered sufficient to provide adequate information for the study objectives.

### 5.2 Definition of analysis sets

#### 5.2.1 Full analysis set

The Full Analysis Set (FAS) will consist of all subjects who have been randomised and used at least one of the IPs and who has at least one post-baseline assessment of data.

#### 5.2.2 Pharmacokinetic analysis set

The Pharmacokinetic analysis set (PKAS) will consist of all subjects who used at last one of the IPs and provided an evaluable plasma concentration profile and who have no AEs or protocol deviations judged to affect the PK analysis. Individual PK values may be excluded from the analysis as specified in the SAP. The PKAS will be used as the per protocol analysis set.

#### 5.2.3 Use of analysis set

The use of the analysis sets/populations is indicated for each table/figure/listing under statistical output layout .

#### **5.3** Definition of baseline

The baseline measurement is defined as the latest measurement prior to first IP exposure of each treatment period of the IP.

### 5.4 Output rounding principles

Generally, no rounding of data will be done prior to calculating statistics. However, if reported data contains more than 8 significant digits it will be rounded to 8 significant digits in the database.

In statistical output and descriptive summaries, the following principles will be followed:

- 3 significant digits will be used for PK and similar parameters.
- 2 significant digits will be used for percentages (for example relative change from baseline).
- p-values and similar statistical output will be presented using 4 decimal points.
- All descriptive summaries of numerical data (e.g. mean, SD etc.) will be presented with one extra decimal compared to reported input data.


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



### 5.5 Significance level

When testing equivalence (as for the primary endpoint), a significance level of 10% will be used ( $\alpha$ =0.10). All other hypothesis testing (when not testing equivalence) will use a 5% significance level ( $\alpha$ =0.05).

### 5.6 Multiple comparisons/multiplicity

No adjustment for multiple comparison/multiplicity will be performed. All significant findings will be reviewed for medical relevance.

### 5.7 Handling of dropouts, missing data and outliers

Outliers will be included in summary tables and listings and will not be handled separately in any analyses. Generally, no imputation of data will be performed. However, clinical safety laboratory parameters that are outside the detection limit, will be replaced with the detection limit when calculating statistics. Also, when calculating statistics for PK plasma concentrations, concentrations under LLOQ will be replaced with LLOQ if more than 50% of the values for a given time point is above LLOQ. Otherwise, no statistics will be calculated for that time point. For imputation of PK plasma concentration under LLOQ with the purpose of calculating PK parameters, see section 6 below.

#### **6** PHARMACOKINETIC ANALYSIS

The PK analysis will be based on the PKAS and performed by CTC. The PK parameters will be calculated by Non-Compartmental Analysis (NCA) using the software Phoenix WinNonlin® version 8.1 or later (Certara, U.S.A).

The following non-compartmental PK parameters will be determined for each IP use:

- C<sub>max</sub> The maximum observed plasma concentration
- AUC<sub>t</sub>-The area under the plasma concentration versus time curve (AUC) from timepoint 0 to t, where t represents the timepoint of the last detectable plasma concentration
- T<sub>max</sub> Time to C<sub>max</sub>
- C<sub>last</sub> The last observed plasma concentration
- AUC<sub>0-90</sub> AUC from timepoint 0 to 90 minutes
- AUC<sub>inf</sub> AUC from timepoint 0 extrapolated to infinity using lambda<sub>z</sub>
- $T_{1/2}$  The terminal plasma elimination half-life

Also, the PK parameters normalised by dose will be calculated.

Analysis will be based on the actual sampling times recorded during the study. of calculating PK parameters, concentrations below lower limit of quantification (LLOQ) occurring before  $C_{max}$  will be treated as zero. Concentrations below LLOQ occurring after  $C_{max}$  will be omitted from the analysis.

 $C_{max}$ ,  $T_{max}$  and  $C_{last}$  will be derived from the observed plasma concentration data. AUC will be assessed by integration of the plasma concentration vs time curve using linear interpolation for increasing plasma levels and logarithmic interpolation for decreasing plasma levels


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



(Linear Up-Log Down method). AUC<sub>t</sub> will be calculated from time 0 to the time t of the last detectable plasma concentration. AUC<sub>0-90</sub> is the AUC truncated at 90 min. If there is no actual sampling time point at 90 min, the concentration at 90 min will be determined by interpolation between the surrounding actual sampling points (according to linear up, log down principles). For AUC<sub>inf</sub> the area will be calculated to the last timepoint showing a measurable plasma concentration and then extrapolated to infinity using the concentration in the last quantifiable sample and lambda<sub>z</sub>. T<sub>½</sub> will be calculated by ln 2 / lambda<sub>z</sub>.

Lambda<sub>z</sub>, the first order rate constant associated with the terminal portion of the curve will be determined by lin-logarithmic regression of the terminal elimination phase of individual plasma concentration vs time curves. Determination of lambda<sub>z</sub> requires identification of a sufficiently linear terminal phase (as determined by visual inspection of the lin-log plasma concentration vs time plot with the regression line) consisting of at least 3 terminal concentration values (not including  $C_{max}$ ). If this is not achieved, lambda<sub>z</sub> and its dependent PK parameters will not be reported for that profile. In the following cases, lambda<sub>z</sub> dependent PK parameters will be flagged in listings as potentially unreliable:

- Lambda<sub>z</sub> estimation is based on a period of less than 1.0 times the resulting  $T\frac{1}{2}$ .
- The adjusted R2 value of the regression line is < 0.85.
- The estimated % extrapolated AUC is  $\geq 20\%$  ((AUC<sub>inf</sub> -AUC<sub>t</sub> / AUC<sub>inf</sub>)\*100).

Where plasma nicotine concentrations are above LLOQ immediately prior to product administration (pre-dose sample), PK parameters will also be calculated from baseline adjusted concentrations using a subject's elimination rate constant (lambda<sub>z</sub>) (from the curve during the specific treatment period) and observed pre-dose concentration (considered to have been collected at time 0). Baseline adjustments will be calculated according to the formula:

$$C(t)_{adjusted} = C(t)_{observed} - C(0)e^{-lambdaz(t)}$$

In cases of a generated negative  $C(t)_{adjusted}$ , the value will be replaced with zero.

Where plasma nicotine concentrations are below LLOQ immediately prior to product administration (pre-dose sample), baseline adjusted PK parameters will be considered the same as non-baseline adjusted PK parameters.

For subjects where lambda<sub>z</sub> cannot be calculated, baseline adjusted PK parameters ( $C_{max}$ , AUC<sub>t</sub>,  $T_{max}$ ,  $C_{last}$ , AUC<sub>0-90</sub>, AUC<sub>inf</sub> and  $T_{1/2}$ ) will not be generated and reported. For subjects where lambda<sub>z</sub> can be calculated but where the acceptance criteria for lambda<sub>z</sub> determination have not be fulfilled, baseline adjusted PK parameters will be calculated, but reported PK parameters will then be flagged in listings as potentially unreliable.

In addition to PK parameters specified in the protocol,  $t_{last}$  (the time of Clast),  $AUC_{extr}$ %, lambda<sub>z</sub> and details about lambda<sub>z</sub> determination (adjusted R<sub>2</sub>, span, number of timepoints and lower/ upper timepoints used for lambda<sub>z</sub> calculation) will be presented in the listing section.

If there is a confirmed dosing error during the study, the PK data for that period will only be included in the listings but excluded from descriptive and statistical analyses. In case of missed blood samples, potential impact on PK parameters will be assessed for each individual case. PK parameters with a high degree of uncertainty due to missing samples (e.g. multiple


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



samples missing around  $C_{max}$ ) will be flagged as unreliable in the report and may in rare cases be excluded from summary tables, descriptive statistics, and statistical analysis.

### 7 CLINLCAL DATABASE PROCESSING

#### 7.1 General information

The standards set forth by the Clinical Data Interchange Standards Consortium (CDISC) will be followed. CDISC develops and publishes standards in order to normalise the structure of clinical study data and thereby simplify submissions to and reviews by authorities such as the Food and Drug Administration (FDA). These standards include naming conventions, code lists, and data structure formats.

The study data will be structured into a database model reflecting the Study Data Tabulation Model (SDTM) and be compliant to SDTM Implementation Guide (SDTM-IG) version 3.2. The data used for statistical analysis will be structured to reflect the Analysis Data Model (ADaM) and be compliant to ADaM Implementation Guide (ADaM-IG) version 1.1. Both SDTM and ADaM are data-model standards developed by CDISC, and the versions used are mentioned as preferred versions in the FDA data standards catalogue.

Data values are collected according to, or mapped into, Controlled Terminology (CT) codelists defined by CDISC, whenever possible. The codelists are updated annually at CTC and the latest version available at study start will be used. As per default, CT codelists will be used in all tables, listings, and figures. Custom codelists for test or parameter names will be used if applicable upon Sponsor's request, to align with protocol texts, or to adhere to other standard naming conventions (e.g. PK parameter name "Tmax" will be used instead of the CDISC term "Time of CMAX"). These custom codelists will be mapped in the "Parameter Name" field in the ADaM structure, while the CT will be kept in the SDTM predecessor fields to provide traceability back to CDISC codelists.

#### 7.2 Database modeling of study design

The SDTM study design model contains the following structural components:

**EPOCH**: Study epochs follow a controlled terminology to represent the different study parts (e.g. SCREENING, TREATMENT [X], FOLLOW-UP)

**ELEMENT**: Building blocks used to build up the entire study length for all subjects. Information on ELEMENTs are extracted from the study design and schedule of events in the protocol. ELEMENTs are defined to span the entire study without gaps. One EPOCH may contain one or several ELEMENTs. All ELEMENTs must have transition rules in accordance with the protocol to determine start and end.

**ARM**: Subjects are allocated to study arms depending on the study design, either by randomisation or other allocation processes defined in the study protocol. ARMs are defined as the total number of planned ways a subject can go through the study (unique combination of study ELEMENTs). All ARMs must contain a unique sequence of ELEMENTs.


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



**VISIT**: Study visits are defined as planned timepoints during the study where study data is collected. A visit can be performed in clinic, by off-site contact with study personnel (phone call, video conference or similar), or by subject initiated recordings of data. The visit schedule is extracted from protocol and eCRF design.

Below is a schematic representation of the SDTM study design:



#### 8 STATISTICAL METHODOLOGY

All relevant collected data will be listed. Additional statistical analyses and descriptive summaries are specified below.

### 8.1 Primary endpoint(s) analysis

#### 8.1.1 C<sub>max</sub> and AUC<sub>t</sub>

This section refers to the primary objective 1, endpoint 1.1.

 $C_{max}$  and  $AUC_t$  and baseline adjusted  $C_{max}$  and  $AUC_t$  will be summarised descriptively. Also, log transformed nicotine  $C_{max}$  and  $AUC_t$  estimates will be evaluated separately in a linear mixed-effects analysis of variance model with fixed effects for product and a random effect for subject. The above product differences will be back-transformed to present the ratios of geometric least squares (LS) means coupled with the 90% confidence intervals (CIs). If the CI falls within the range of 0.8-1.25, the corresponding two products are considered equivalent with respect to that comparison.

## 8.1.2 Tables and Figures relating to the primary endpoint(s)

Analysis and output related to the primary endpoint(s) are specified under section statistical output layout. The following tables and figures relate to the primary endpoint(s):

Table 14.4.1 PK parameters (Pharmacokinetic analysis set)

Table 14.4.2 PK parameters – Normalised by dose (Pharmacokinetic analysis set)

**Error!** Reference source not found.


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



### 8.2 Secondary endpoint(s) analysis

### 8.2.1 Definition of endpoint(s)

8.2.1.1 Other Pharmacokinetic parameters  $T_{max}$ ,  $C_{last}$ ,  $AUC_{0-90}$ ,  $AUC_{inf}$  and  $T_{1/2}$  and and baseline adjusted  $T_{max}$ ,  $C_{last}$ ,  $AUC_{0-90}$ ,  $AUC_{inf}$  and  $T_{1/2}$ 

This section refers to the secondary objective 2.1, endpoints 2.1.1.

See Section 6. All PK parameters (and PK parameters normalised by dose) will be summarised descriptively.

### 8.2.1.2 Extracted dose of nicotine

This section refers to the secondary objective 2.2, endpoint 2.2.1.

Content pre-use is calculated by multiplying the mean content of the weight normalised reference samples with the pouch weight of the study pouches. Content post-use is the measured content left in the study pouches post-use. Extracted amount (mg/unit) of nicotine, for each pouch, is calculated as the difference of content pre-use and content post-use, i.e.:

Equation 1

$$(D \times E_i) - F_i$$
  
 $i = 1, ..., N$ 

where *N*=number of study pouches used in analysis

D= Mean content of weight normalised reference samples

 $E_i$  = Weight of the unused pouch

 $F_i$  = Content post-use

D is calculated by:

$$D = \frac{\sum_{j=1}^{M} C_j}{M},$$

where  $C_j = \frac{A_j}{B_j}$  is weight normalised content for reference samples, and  $A_j$ =reference nicotine amount and  $B_i$ =reference weight, j = 1, ..., M. M=Number of reference samples.

Extracted fraction (%) of nicotine, for each pouch i = 1, ..., N, is calculated as the extracted amount divided by the content pre-use, i.e.:

Equation 2

$$\frac{(D \times E_i) - F_i}{D \times E_i}$$

Extracted dose of nicotine will be summarised descriptively and analysed using a Wilcoxon signed rank test to assess differences between IPs.

Pearson correlation coefficients for baseline adjusted AUC<sub>inf</sub>, AUC<sub>t</sub>, baseline adjusted AUC<sub>inf</sub> and baseline adjusted AUC<sub>t</sub>and the derived extracted dose of nicotine (attained via Equation 1 above) will be estimated and presented for each IP, with corresponding p-value.


Protocol Version No: Final v1.0: 21JUN2021

Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



#### 8.2.1.3 Product evaluation scale (PES)

This section refers to the secondary objective 2.3, endpoint 2.3.1.

Each question of the PES will be answered using a 7-point Likert scale. Responses will be presented as the following factor scores: 1 = not at all, 2 = very little, 3 = a little, 4 = moderately, 5 = a lot, 6 = quite a lot, 7 = extremely.

Four multi-item subscales will be derived from the PES categories:

- "Satisfaction" (items 1, 2, 3, and 12)
- "Psychological Reward" (items 4-8)
- "Aversion" (items 9, 10, 16, and 18)
- "Relief" (items 11, 13, 14, 15, and reversed for item 20)

These four multi-item subscales will be summarized descriptively by IP and overall, at applicable assessment timepoints. Single items 17, 19 and 21 will also be summarized in the same way as the multi-item subscales. Also, PES sub-category and total scores will be presented visually with individual and mean figures.

In addition, PES-differences between products on total and sub-category PES score, at each time point, will be analysed using Wilcoxon Rank Sum tests.

#### 8.2.1.4 Product preference scale (PPS)

Park the 1 nauch products in relation to

This section refers to the secondary objective 2.3, endpoint 2.3.1.

PPS will be summarised descriptively by IP. The PPS data collected in the eCRF will therefore be derived so the results will be presented by IP, instead of presented by day (as collected) i.e., derived according to the following:

| Rank the 4 pouch products in relation to each other. | | | | | Rate the 4 poucl preference | n prod | ucts in | order o | f |
|---|---|---|---|---|---|---|---|---|---|
| Study product used at: | Ord | ler of pi | eferenc | e: | Study product: | Pref | ference | result: | |
| Day 1 | 1 | 2 | 3 | 4 | Product A | 1 | 2 | (3) | 4 |
| Day 2 | 1 | 2 | 3 | 4 | Product B | (1) | 2 | 3 | 4 |
| Day 3 | 1 | 2 | 3 | 4 | Product C | 1 | 2 | 3 | 4 |
| Day 4 | 1 | (2) | 3 | 4 | Product D | 1 | 2 | 3 | $\overline{(4)}$ |

Note: this is just an illustrative example with made up subject evaluations, to explain the data derivation. The table layout for PPS can be found in Table 14.2.3 Products preference scale (PPS) (Full analysis set)

#### 8.2.1.5 *Urge to use questionnaire*

This section refers to the secondary objective 2.3, endpoint 2.3.1.

The answer from the Urge to use questionnaire is graded on a Visual Analogue Scale (VAS) from 0-100 mm, where 0 is "No urge at all" and 100 is "extreme urge".

The following parameters will be calculated for the urge to use assessments:

- E<sub>max</sub> The maximum change from baseline VAS score (VAS<sub>pre-use</sub> VAS<sub>post-use</sub>).
- $T_{Emax}$  Time of the  $E_{max}$ . If the maximum value occurs at more than one time point,  $T_{\text{Emax}}$  will be defined as the first time point with this value.


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



• AUEC<sub>0-120</sub> - The area under the change from baseline VAS score versus time curve from time 0 to 120 minutes, calculated using the linear trapezoidal method with linear interpolation using actual sample times.

Responses and the derived parameters mentioned above will be summarized by IP and overall using descriptive statistics, including change from baseline. Also, urge to use questionnaire (VAS score) will be presented visually with individual and mean figures.

#### 8.2.1.6 Adverse events

This section refers to the secondary objective 2.4, endpoint 2.4.1.

An overview of all AEs, including SAEs, intensity, relationship to IP, and deaths will be presented by IP and overall. Incidence of AEs and SAEs will also be summarised by SOC and PT by IP and overall. For both summaries, any AE that occurred during follow-up, will be presented separately (in an own column, in the same tables).

## 8.2.1.7 Safety laboratory analyses

This section refers to the secondary objective 2.4, endpoint 2.4.2.

Clinical laboratory data will be summarised by IP with absolute and percent change from baseline.

### 8.2.1.8 Vital signs

This section refers to the secondary objective 2.4, endpoint 2.4.2.

Vital signs (systolic/diastolic blood pressure and pulse) will be summarised by IP. Data will be presented with absolute and percent change from baseline.

#### 8.2.1.9 12-lead ECG

This section refers to the secondary objective 2.4, endpoint 2.4.2.

All ECGs will be categorised as "normal", "abnormal, not clinically significant", or "abnormal, clinically significant" (as judged by the Investigator) and summarised by IP using frequency tables.

#### 8.2.2 Tables and Figures relating to the secondary endpoint(s)

Analysis and output related to the secondary endpoint(s) are specified under section statistical output layout. The following tables and figures relate to the secondary endpoint(s):

Table 14.2.1 Products evaluation scale (PES) (Full analysis set)

Table 14.2.2 Products evaluation scale (PES) – Wilcoxon Rank Sum tests comparison of treatments (Full analysis set)

Table 14.2.3 Products preference scale (PPS) (Full analysis set)

Table 14.2.4 Urge to use questionnaire (Full analysis set)

Table 14.2.5 Urge to use questionnaire – Treatment comparisions (Full analysis set)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



Table 14.3.1 Overview of adverse events (Full analysis set)

Table 14.3.2 Adverse events by system organ class and preferred term (Full analysis set)

Table 14.3.3 Safety laboratory measurements - clinical chemistry (Full analysis set)

Table 14.3.4 Safety laboratory interpretations - clinical chemistry (Full analysis set)

Table 14.3.5 Safety laboratory measurements - haematology (Full analysis set)

Table 14.3.6 Safety laboratory interpretations - haematology (Full analysis set)

Table 14.3.7 Vital signs measurements (Full analysis set)

Table 14.3.8 Vital signs interpretations (Full analysis set)

Table 14.3.9 ECG measurements (Full analysis set)

Table 14.3.10 ECG interpretations (Full analysis set)

Table 14.3.11 Physical examinations (Full analysis set)

Table 14.3.12 Physical examinations interpretations (Full analysis set)

Table 14.3.13 Plasma concentrations (Pharmacokinetic analysis set)

Table 14.4.1 PK parameters (Pharmacokinetic analysis set)

Table 14.4.2 PK parameters – Normalised by dose (Pharmacokinetic analysis set)

8.2.2.1.1.1 Table 14.4.3 PK parameters – Treatment comparisons (Pharmacokinetic analysis set)

Table 14.4.4 Extracted dose of nicotine - normalised by weight and relative amount (Full analysis set)

Table 14.4.5 Extracted dose of nicotine – Wilcoxon Signed Rank tests comparison of treatments (Pharmacokinetic analysis set)

Table 14.4.6 Extracted dose of nicotine – Pearson correlations to PK parameters (Pharmacokinetic analysis set)

Figure 14.2.1 Products evaluation scale (PES) sub-category and total scores individual graphs (Full analysis set)

Figure 14.2.2 Products evaluation scale (PES) sub-category and total scores mean graphs (Full analysis set)

Figure 14.2.3 Urge to use (VAS score) individual graphs (Full analysis set)

Figure 14.2.4 Urge to use (VAS Score) mean graphs (Full analysis set)

Figure 14.4.1 Individual plasma concentrations over time (lin-log) (Pharmacokinetic analysis set)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



Figure 14.4.2 Individual plasma concentrations over time (lin-lin) (Pharmacokinetic analysis set)

Figure 14.4.3 Mean plasma concentrations over time (lin-log) (Pharmacokinetic analysis set)

Figure 14.4.4 Mean plasma concentrations over time (lin-lin) (Pharmacokinetic analysis set)

### 8.3 Tertiary/exploratory endpoint(s) analysis

NA

## 8.4 Other data analysis/presentation

- 8.4.1 Demographics and baseline characteristics Descriptive statistics for demographics, physical examinations, weight and height will be presented by sequence.
- 8.4.2 Medical/surgical history and prior/concomitant medication Medical/surgical history will be presented by system-organ-class (SOC) and preferred term (PT). Prior/concomitant medications will be presented by ATC level 3 and 5. Medical/surgical history and prior medications will be presented overall by descriptive statistics and listings. Concomitant medications will be presented by sequence.

In addition to the primary and secondary endpoint(s) described above, the following tables and figures will be produced:

Table 14.1.1 Baseline characteristics and demographics (Full analysis set)

Table 14.1.2 Subject disposition (all subjects)

Table 14.1.3 Medical history events by system organ class and preferred term (Full analysis set)

Table 14.1.4 Concomitant medications by ATC levels 3 and 5 (Full analysis set)

Table 14.1.5 Prior medications by ATC levels 3 and 5 (Full analysis set)

### 8.5 Interim analysis

NA

#### 9 CHANGES FROM THE CSP

### 9.1 Changes of product comparisons for primary analysis

In the protocol (Synopsis and Section 17.5) it was stated that the primary objective will be examined by the following statistical comparisons for AUC and C<sub>max</sub>:

o Product A versus Product B, C and D, respectively


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



- o Product B versus Product C and D, respectively
- o Product C versus Product D

Instead, the primary objective will be examined by the following statistical comparisons for  $AUC_t$  and  $C_{max}$ :

- o Product A does not significantly differ from Product D
- o Product B does not significantly differ from Product D
- o Product C does not significantly differ from Product D

The reason for the change is that the test products are Products A-C and the Comparator product is Product D, so there is no need for multiple comparisons.

## 9.2 Changes of fixed effects for primary analysis

In the protocol (Synopsis and Section 17.5) it was stated that the linear mixed-effects model for the primary analysis should include fixed effects for period, sequence, and product, and a random effect for subject. The fixed effects for period and sequence will be removed for the statistical analysis. The subjects will be allowed to use their own nicotine containing products ad lib after the 8-hour timepoint until 10 pm. Hence, keeping period and sequence in the model adds no extra value to the analysis.

### 9.3 Change of analysis method for Urge to use questionnaire for secondary analysis

In the protocol it was stated that the same statistical method as described for the PK analysis will be used to compare Urge to use parameters. Instead, change from baseline will be evaluated descriptively for each IP.

#### 10 STATISTICAL DELIVERABLES

The following documents will be delivered:

- SAP
- Statistical analyses, summary tables, listings and figures as described under section 14
- Clinical study database delivered as a SAS-export file.

#### 11 SOFTWARE

All statistical analyses will be performed using SAS Version 9.4 (SAS institute, Cary, NC).


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



## **12** APPROVAL

| Issued by: | |
|-----------------------------|------|
| Responsible Biostatistician | Date |
| CTC Representative | |
| Approved by: | |
| PP | |


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021



## 13 SUPPORTIVE DOCUMENTATION

## 13.1 Appendix 1 – list of abbreviations

| Abbreviation of term | Explanation |
|----------------------|---------------------------------------------------|
| ADaM | Analytical Data Model |
| AE | Adverse event |
| ATC | Anatomical-therapeutic-chemical |
| APTT | Activated partial thromboplastin time |
| CDISC | Clinical Data Interchange Standards<br>Consortium |
| CF | Clean file |
| CI | Confidence interval |
| CRF | Case report form |
| CSP | Clinical study protocol |
| ECG | Electrocardiogram |
| FAS | Full analysis set |
| IP | Investigational product |
| LLOQ | Lower level of quantification |
| Max | Maximum |
| MedDRA | Medical Dictionary for Regulatory Affairs |
| Min | Minimum |
| NA | Not applicable |
| OND | Oral nicotine delivery |
| PES | Product evaluation scale |
| PPS | Product preference scale |
| PPS | Per protocol set |
| PT | Preferred term |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS | Statistical analysis system |
| SD | Standard deviation |


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

### 14 STATISTICAL OUTPUT LAYOUT

Placeholder descriptions like "GROUP 1", "Treatment A", "ELEMENT 1" etc. below should be replaced by appropriate.

## 14.1 Template tables

Template tables will be adjusted as needed depending on the collected data. For example, if there is only one will be dropped and the Result category column will also be dropped, as there is no second time point for who baseline to. Optional columns will not be included in specific output unless explicitly stated.

22 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

## Template table A Descriptive statistic table – continuous variables

| | | | | GROUP 1 | GR |
|---|---|---|---|---|---|
| Assessment (unit) | Result category | Assessment timepoint | | | 1 |
| [Parameter 1] (unit) | Measured value | [Assessment timepoint 1] | n | x | х |
| | | | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.x |
| | | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx (x.x |
| | | [Assessment timepoint 2] | n | x | X |
| | | | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.x |
| | | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx (x.x |
| | Absolute change from baseline | [Assessment timepoint 2] | n | x | X |
| | | | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.x |
| | | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx (x.x |
| | Relative change from baseline (%) | [Assessment timepoint 2] | n | x | x |
| | | | Mean (SD) | x.x (x.x) | x.xxx (x.x |
| | | | Median (Min, Max) | x.x (x, x) | x.xxx (x.x |

Data based on [ANALYSIS SET]. Baseline at [Assessment timepoint 1]. ND: Not defined - no evaluable observations missing observations. NC: Not calculated - number of non-missing observations less than 3 [STUDYID] [DOMAIN]: [PARAMETER CATEGORY], SAS program: descriptive\_stat\_tables.sas. Run by: [USERNAME], [TIME]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

## Template table B Descriptive statistic table – discrete variables

| | | | | GROUP 1 | GROUP 2 | [Tota |
|---|---|---|---|---|---|---|
| Assessment | Assessment timepoint | Result | | | | |
| [Parameter 1] | [Assessment timepoint 1] | [RESULT 1] | X | (x.x%)/X | x(x.x%)/X | x(x.x%)/. |
| | | [RESULT 2] | X | (x.x%)/X | x(x.x%)/X | x(x.x%)/. |
| | [Assessment timepoint 2] | [RESULT 1] | X | (x.x%)/X | x(x.x%)/X | x(x.x%)/. |
| | | [RESULT 2] | X | (x.x%)/X | x(x.x%)/X | x(x.x%)/. |

Data based on [ANALYSIS SET].

[STUDYID] [DOMAIN]: [PARAMETER CATEGORY], SAS program: descriptive\_stat\_tables.sas. Run by: [USERNAME], [TIME


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 24 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

## 14.2 Template figures

Template figures will be adjusted as needed depending on the collected data.

Template figure A Subject measurements over time by treatment figure



Data based on [ANALYSIS SET].
[STUDYID] [DOMAIN]: [PARAMETER CATEGORY], SAS program: [PROGRAM NAME]. Run by: [USERNAME], [TIMESTAMP]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

## Template figure B Treatment measurements over time by subject figure



Data based on [ANALYSIS SET].
[STUDYID] [DOMAIN]: [PARAMETER CATEGORY], SAS program: [PROGRAM NAME]. Run by: [USERNAME], [TIMESTAMP]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Template figure C Measurements over time by treatment with confidence interval bars figure



Data based on [ANALYSIS SET]. Confidence intervals calculated from a normal distribution.
[STUDYID] [DOMAIN]: [PARAMETER CATEGORY], SAS program: [PROGRAM NAME]. Run by: [USERNAME], [TIMESTAMP]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

## **14.3 Tables**

Table 14.1.1 Baseline characteristics and demographics (Full analysis set)

| | | A:B:C:D<br>(N=X) | B:C:D:A<br>(N=X) | C:D:A:B<br>(N=X) |
|---|---|---|---|---|
| Age (years) | n/nmiss | x/x | x/x | x/x |
| | Mean (SD) | x.x (x.x) | x.x(x.x) | x.x (x.x) |
| | Median (Min, Max) | x.x(x, x) | x.x(x, x) | x.x(x, x) |
| Body Mass Index (kg/m²) | n/nmiss | x/x | x/x | x/x |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx (x.x, 2 |
| Height (cm) | n/nmiss | x/x | x/x | x/x |
| | Mean (SD) | x.x (x.x) | x.x(x.x) | x.x(x.x) |
| | Median (Min, Max) | x.x(x, x) | x.x(x, x) | x.x(x, x) |
| Weight (kg) | n/nmiss | x/x | x/x | x/x |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx (x.x, y |
| Sex | Female | x (x.x%) | x (x.x%) | x (x.x%) |
| | Male | x (x.x%) | x (x.x%) | x (x.x%) |
| Ethnicity | Hispanic Or Latino | x (x.x%) | x (x.x%) | x (x.x%) |
| | Not Hispanic Or Latino | x (x.x%) | x (x.x%) | x (x.x%) |
| | Not Reported | x (x.x%) | x (x.x%) | x (x.x%) |
| | Unknown | x (x.x%) | x (x.x%) | x (x.x%) |
| Race | American Indian Or Alaska Native | x (x.x%) | x (x.x%) | x (x.x%) |
| | Asian | x (x.x%) | x (x.x%) | x (x.x%) |
| | Black or African American | x (x.x%) | x (x.x%) | x (x.x%) |
| | Native Hawaiian or other Pacific Islander | x (x.x%) | x (x.x%) | x (x.x%) |


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

| | A:B:C:D | B:C:D:A | C:D:A:B |
|-------|----------|----------|----------|
| | (N=X) | (N=X) | (N=X) |
| White | x (x.x%) | x (x.x%) | x (x.x%) |

[STUDYID] Summarised demographics data.

Data based on the [Full analysis set].

SAS program: summary\_demographics.sas. Run by: [USERNAME], [TIMESTAMP]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 29 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.1.2 Subject disposition (all subjects)

| | Total |
|-------------------------------|-------|
| Screened subjects | X |
| Withdrawn prior to dose | X |
| Withdrawal reason x | X |
| Withdrawal reason x | X |
| Withdrawal reason x | X |
| Included subjects | X |
| A:B:C:D | X |
| B:C:D:A | X |
| C:D:A:B | X |
| D:A:B:C | X |
| Withdrawn subjects | X |
| Withdrawal reason x | X |
| Withdrawal reason x | X |
| Withdrawal reason x | X |
| Completed subjects | X |
| Included in full analysis set | X |
| Included in PK analysis set | X |
| Subjects at Screening | X |
| Subjects at In-Clinic | X |
| Subjects at Phone Call | X |

[STUDYID] Disposition, SAS program: disposition.sas. Run by: [USERNAME], [TIMESTAMP]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.1.3 Medical history events by system organ class and preferred term (Full analysis set)

| | Total<br>N=X | |
|--------------------------------------|--------------|---|
| System organ class<br>Preferred term | n(%) | m |
| Total | x(x.x%) | X |
| SOC 1 | x(x.x%) | X |
| SOC 1 PT 1 | x(x.x%) | X |
| SOC 1 PT 2 | x(x.x%) | X |
| SOC 1 PT 3 | x(x.x%) | X |
| SOC 2 | x(x.x%) | X |
| SOC 2 PT 1 | x(x.x%) | X |
| SOC 2 PT 2 | x(x.x%) | x |

n, number of subjects; m, number of events

Percentages are based on the number of subjects in the treatment period included in the [Full analysis set]

[STUDYID] Medical history events by system organ class and preferred term, [analysis set], SAS program: mh\_s

[USERNAME], [TIMESTAMP]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.1.4 Concomitant medications by ATC levels 3 and 5 (Full analysis set)

| | A:B:C:D<br>N=X | B:C:D:A<br>N=X | C:D:A:B<br>N=X |
|---|---|---|---|
| ATC Name Level 3<br>ATC Name Level 5 | n(%) m | | n n(%) m |
| Total | x(x%) x | x(x%) | x x(x%) x |
| | x(x%) X | $x(x^{0/0})$ | X = x(x%) = X |

n, number of subjects; m, number of events

Percentages are based on the number of subjects in the full analysis set

[STUDYID] Medical history events by system organ class and preferred term, [Full analysis set], SAS program:

by: [USERNAME],] [TIMESTAMP]

Table 14.1.5 Prior medications by ATC levels 3 and 5 (Full analysis set)

| Total | x(x%)<br>x(x%) | x<br>X |
|--------------------------------------|----------------|--------|
| ATC Name Level 3<br>ATC Name Level 5 | n(%) | m |
| | Total<br>N=X | |

n, number of subjects; m, number of events

Percentages are based on the number of subjects in the full analysis set

[STUDYID] Medical history events by system organ class and preferred term, [Full analysis set], SAS program:

by: [USERNAME], [TIMESTAMP]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 32 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.2.1 Products evaluation scale (PES) (Full analysis set)

[Note to programmer: multi-items and single-items are defined in Section 8.2.1.3]

| | | | A | В | C |
|---|---|---|---|---|---|
| Assessment | Assessment timepoint | Result | | | |
| Satisfaction (multi-item 1) | [Assessment timepoint 1] | Not at all (1) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| | | Very little (2) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| | | | | ••• | ••• |
| | [Assessment timepoint 2] | Not at all (1) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| | | Very little (2) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| Psychological Reward (multi-item 2) | [Assessment timepoint 1] | Not at all (1) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| (main tem 2) | | Very little (2) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| | [Assessment timepoint 2] | Not at all (1) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| | | Very little (2) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| | | | | ••• | |
| Was it easy to use? (single-<br>item 17) | [Assessment timepoint 1] | Not at all (1) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| ., | | Very little (2) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| | [Assessment timepoint 2] | Not at all (1) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |
| | | Very little (2) | x(x.x%)/X | x(x.x%)/X | x(x.x%)/X |


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.2.2 Products evaluation scale (PES) – Wilcoxon Rank Sum tests comparison of treatment

| Question multi-item sub-<br>category | Assessment timepoint | Test product | Reference product | 95%<br>CI<br>lower<br>bound | Estimated difference | 95%<br>CI<br>upper<br>bound | p-value |
|---|---|---|---|---|---|---|---|
| Satisfaction | [Assessment timepoint 1] | Product A | Product D | x.xx | x.xxxx | x.xxx | x.xxxx |
| | | Product B | Product D | x.xx | x.xxxx | x.xxx | x.xxxx |
| | | Product C | Product D | x.xx | x.xxxx | x.xxx | x.xxxx |
| Psychological Reward | [Assessment timepoint 1] | Product A | Product D | x.xx | x.xxxx | x.xxx | x.xxxx |
| | | Product B | Product D | x.xx | x.xxxx | x.xxx | x.xxxx |
| | | ••• | | | | | |


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 34 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

### Table 14.2.3 Products preference scale (PPS) (Full analysis set)

[Note to programmer: PPS will be summarised descriptively by IP. The PPS data collected in the eCRF will therefore be derived so of presented by day (as collected), see Section 8.2.1.4]

| Product preference order | Result | Total |
|--------------------------|--------|-----------|
| Product A | 1 | x(x.x%)/X |
| | 2 | x(x.x%)/X |
| | 3 | x(x.x%)/X |
| | 4 | x(x.x%)/X |
| Product B | 1 | x(x.x%)/X |
| | 2 | x(x.x%)/X |
| | 3 | x(x.x%)/X |
| | 4 | x(x.x%)/X |
| Product C | 1 | x(x.x%)/X |
| | 2 | x(x.x%)/X |
| | 3 | x(x.x%)/X |
| | 4 | x(x.x%)/X |
| Product D | 1 | x(x.x%)/X |
| | 2 | x(x.x%)/X |
| | 3 | x(x.x%)/X |
| | 4 | x(x.x%)/X |

Data based on [ANALYSIS SET].

Results are presented as n(%)/N, where N is the total number of observations at that specific timepoint. Order products: 1 = most preferred product, 4 = least preferred product.
[STUDYID] [DOMAIN]: [PARAMETER CATEGORY], SAS program: descriptive\_stat\_tables.sas. Run by: [USERNAME], [TIME


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.2.4 Urge to use questionnaire (Full analysis set)

| | | | A | В | C | |
|---|---|---|---|---|---|---|
| Assessment (unit) | Assessment timepoint | | | | | |
| Urge to use (unit) | [Assessment | n | x | x | X | х |
| | timepoint 1] | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | X.XX |
| | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx (x.xx, x.xx) | x.xxx (x.xx, x.xx) | X.XX |
| | [Assessment | n | x | x | x | x |
| | timepoint 2] | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | X.XX |
| | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx (x.xx, x.xx) | x.xxx (x.xx, x.xx) | x.xx |
| Emax (unit) | [Assessment | n | x | x | x | x |
| | timepoint 1] | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | X.XX |
| | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx(x.xx, x.xx) | x.xxx (x.xx, x.xx) | X.XX |
| | [Assessment timepoint 2] | n | x | X | X | x |
| | штерет 2, | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | X.XX |
| | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx(x.xx, x.xx) | x.xxx(x.xx, x.xx) | X.XX |
| TEmax (unit) | [Assessment | n | x | X | X | x |
| | timepoint 1] | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | X.XX |
| | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx(x.xx, x.xx) | x.xxx(x.xx, x.xx) | X.XX |
| | [Assessment timepoint 2] | n | x | X | X | X |
| | 1 | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | X.XX |
| | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx(x.xx, x.xx) | x.xxx(x.xx, x.xx) | X.XX |
| $AUEC_{0-120}$ (unit) | [Assessment timepoint 1] | n | x | X | X | X |
| | | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xx |
| | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx(x.xx, x.xx) | x.xxx(x.xx, x.xx) | X.XX |
| | | | | | | , |


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021

Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

| | | | A | В | C | |
|---|---|---|---|---|---|---|
| Assessment (unit) | Assessment timepoint | | | | | |
| | [Assessment timepoint 2] | n | x | X | X | х |
| | timepoint 2 <sub>1</sub> | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | X.XX |
| | | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx(x.xx, x.xx) | x.xxx (x.xx, x.xx) | X.XX |

Table 14.2.5 Urge to use questionnaire – Treatment comparisions (Full analysis set)

| Assessment (unit) | Test formulation | Reference formulation | 90%<br>CI<br>lower<br>bound | Ratio of<br>geometric<br>LSMeans | 1.1 | p-value |
|---|---|---|---|---|---|---|
| Emax (unit) | A | D | X.XXX | x.xxxx | x.xxx | X.XXXX |
| | В | D | X.XXX | x.xxxx | x.xxx | X.XXXX |
| | C | D | X.XXX | x.xxxx | x.xxx | X.XXXX |
| TEmax (unit) | A | D | X.XXX | x.xxxx | x.xxx | X.XXXX |
| | В | D | x.xxx | x.xxxx | x.xxx | X.XXXX |
| | C | D | X.XXX | x.xxxx | x.xxx | x.xxxx |

Data based on PK analysis set. Pairwise treatment comparisons are based on a repeated measurement mixed model model has p-value of x.xxxx. [STUDYID] [Full analysis set], SAS program: [PROGRAM NAME]. Run by: [USERNAME],


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 37 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.3.1 Overview of adverse events (Full analysis set)

| | A<br>N=X | | B<br>N=X | | C<br>N=X | | D<br>N=X | | Follow-U<br>N=X | Jp | Total<br>N=X | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n(%) | m | n(%) | m | n(%) | m | n(%) | m | n(%) | m | n(%) | m |
| Any AE | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | x |
| Any SAE | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Any AE leading to withdrawal | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Any AE leading to death | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Causality | | | | | | | | | | | | |
| Unlikely Related | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Possibly Related | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Probably Related | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Severity | | | | | | | | | | | | |
| Mild | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Moderate | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Severe | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Life-threatening | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X |
| Death | x(x.x%) | x | x(x.x%) | X | x(x.x%) | X | x(x.x%) | x | x(x.x%) | X | x(x.x%) | X |

 $<sup>\</sup>ensuremath{\text{n,}}$  number of subjects;  $\ensuremath{\text{m,}}$  number of events

Percentages are based on the number of subjects in the treatment period included in the [Full analysis set]. Adverse events that occurred during screening are omitted from summary.

[STUDYID] Overview of adverse events, [analysis set], SAS program: ae\_summary\_tables.sas. Run by: [USERNAME],


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.3.2 Adverse events by system organ class and preferred term (Full analysis set)

| | A<br>N=X | | B<br>N=X | | C<br>N=X | | D<br>N=X | | Follow-U<br>N=X |
|---|---|---|---|---|---|---|---|---|---|
| System organ class<br>Preferred term | n(%) | m | n(%) | m | n(%) | m | n(%) | m | n(%) |
| SOC 1s | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | x | x(x.x%) |
| SOC 1 PT 1 | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) |
| SOC 1 PT 2 | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) |
| SOC 1 PT 3 | x(x.x%) | x | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) |
| SOC 2 | x(x.x%) | x | x(x.x%) | X | x(x.x%) | X | x(x.x%) | x | x(x.x%) |
| SOC 2 PT 1 | x(x.x%) | x | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) |
| SOC 2 PT 2 | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) | X | x(x.x%) |

n, number of subjects; m, number of events

Percentages are based on the number of subjects in the treatment period included in the Full analysis set Adverse events that occurred during screening are omitted from summary.

[STUDYID] Adverse events by system organ class and preferred term, [analysis set], SAS program: ae\_summary\_by [TIMESTAMP]

39 (49)


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.3.3 Safety laboratory measurements - clinical chemistry (Full analysis set)

#### See appendix

Template table A Descriptive statistic table – continuous variables

[Note to programmer: Clinical laboratory data will be summarised by IP with absolute and percent change from baseline]

Table 14.3.4 Safety laboratory interpretations - clinical chemistry (Full analysis set)

# See appendix

Template table B Descriptive statistic table – discrete variables..

Table 14.3.5 Safety laboratory measurements - haematology (Full analysis set)

#### See appendix

Template table A Descriptive statistic table – continuous variables

[Note to programmer: Clinical laboratory data will be summarised by IP with absolute and percent change from baseline]

Table 14.3.6 Safety laboratory interpretations - haematology (Full analysis set)

### See appendix

Template table B Descriptive statistic table – discrete variables..

Table 14.3.7 Vital signs measurements (Full analysis set)

### See appendix

Template table A Descriptive statistic table – continuous variables. Include all parameters except those include [Note to programmer: Vital signs will be summarised by IP with absolute and percent change from baseline]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 40 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.3.8 Vital signs interpretations (Full analysis set)

See appendix

Template table B Descriptive statistic table – discrete variables. Include all parameters except those included

Table 14.3.9 ECG measurements (Full analysis set)

See appendix

Template table A Descriptive statistic table – continuous variables

Table 14.3.10 ECG interpretations (Full analysis set)

See appendix

Template table B Descriptive statistic table – discrete variables

Table 14.3.11 Physical examinations (Full analysis set)

See appendix

Template table B Descriptive statistic table – discrete variables

Table 14.3.12 Physical examinations interpretations (Full analysis set)

See appendix

Template table B Descriptive statistic table – discrete variables

Table 14.3.13 Plasma concentrations (Pharmacokinetic analysis set)

See appendix

Template table A Descriptive statistic table – continuous variables


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 41 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

## Table 14.4.1 PK parameters (Pharmacokinetic analysis set)

## See appendix

Template table A Descriptive statistic table – continuous variables.

PK parameters to be included in the table (in the following order):

- Non- baseline adjusted:  $T_{max}$ ,  $C_{max}$ ,  $AUC_{0-90}$ ,  $AUC_t$ ,  $AUC_{inf}$ ,  $C_{last}$  and  $T_{1/2}$ .
- Baseline adjusted: T<sub>max</sub>, C<sub>max</sub>, AUC<sub>0-90</sub>, AUC<sub>t</sub>, AUC<sub>inf</sub>, C<sub>last</sub> and T<sub>1/2</sub>.

# Table 14.4.2 PK parameters – Normalised by dose (Pharmacokinetic analysis set)

# See appendix

Template table A Descriptive statistic table – continuous variables.

Table 14.4.3 PK parameters – Treatment comparisons (Pharmacokinetic analysis set)

| Assessment (unit) | Test formulation | Reference<br>formulation | 90%<br>CI<br>lower<br>bound | Ratio of<br>geometric<br>LSMeans | 90%<br>CI<br>upper<br>bound | p-value |
|---|---|---|---|---|---|---|
| AUCt (unit) | A | D | x.xxx | x.xxxx | x.xxx | X.XXXX |
| | В | D | X.XXX | x.xxxx | x.xxx | X.XXXX |
| | C | D | X.XXX | x.xxxx | x.xxx | X.XXXX |
| Cmax (unit) | A | D | X.XXX | x.xxxx | x.xxx | X.XXXX |
| | В | D | X.XXX | x.xxxx | x.xxx | X.XXXX |
| | C | D | x.xxx | x.xxxx | x.xxx | X.XXXX |

Data based on PK analysis set. Pairwise treatment comparisons are based on a repeated measurement mixed model model has p-value of x.xxxx. [STUDYID], [PK analysis set], SAS program: [PROGRAM NAME]. Run by: [USERNAME],


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.4.4 Extracted dose of nicotine - normalised by weight and relative amount (Full analysis

[Note to programmer: Derivations in Section 8.2.1.2]

| | | A | В | C | D |
|---|---|---|---|---|---|
| Assessment (unit) | | | | | |
| NICOTINE (mg/pouch) | n | X | X | X | x |
| | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) |
| | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx(x.xx, x.xx) | x.xxx (x.xx, x.xx) | x.xxx (x.xx, x.xx) |
| NICOTINE (%) | n | x | x | X | x |
| | Mean (SD) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) | x.xxx (x.xxx) |
| | Median (Min, Max) | x.xxx (x.xx, x.xx) | x.xxx(x.xx, x.xx) | x.xxx (x.xx, x.xx) | x.xxx (x.xx, x.xx) |

Data based on Full analysis set.[STUDYID] Adverse events by system organ class and preferred term, [analysis Run by: [USERNAME], [TIMESTAMP]

Table 14.4.5 Extracted dose of nicotine – Wilcoxon Signed Rank tests comparison of treatments

| Parameter (unit) | Test product | Reference product | 95%<br>CI<br>lower<br>bound | Estimated difference | | p-value |
|---|---|---|---|---|---|---|
| NICOTINE (mg/pouch) | A | D | X.XX | x.xxxx | x.xxx | x.xxxx |
| | В | D | X.XX | x.xxxx | x.xxx | X.XXXX |
| | C | D | | | | |
| NICOTINE (%) | A | D | X.XX | x.xxxx | x.xxx | x.xxxx |
| | В | D | x.xx | x.xxxx | x.xxx | x.xxxx |

Data based on PK analysis set.[STUDYID], SAS program: [PROGRAM NAME]. Run by: [USERNAME], [TIMESTAMP]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 43 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Table 14.4.6 Extracted dose of nicotine – Pearson correlations to PK parameters (Pharmacokineti

| PK Parameter (unit) | Extracted dose of nicotine (mg/unit) for Product | Pearson correlation | p-value |
|---|---|---|---|
| Baseline-adjusted AUC <sub>inf</sub> | A | X.XXX | x.xxxx |
| Baseline-adjusted AUC <sub>inf</sub> | В | x.xxx | x.xxxx |
| | ••• | | |

Correlations close to 1 indicates a strong correlation. Data based on PK analysis set.[STUDYID], SAS program: [TIMESTAMP]


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 44 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

### 14.4Figures

Figure 14.2.1 Products evaluation scale (PES) sub-category and total scores individual graphs (Fu

See appendix

Template figure B Treatment measurements over time by subject figure

Figure 14.2.2 Products evaluation scale (PES) sub-category and total scores mean graphs (Full and

See appendix Template figure C Measurements over time by treatment with confidence interval bars figure

Figure 14.2.3 Urge to use (VAS score) individual graphs (Full analysis set)

See appendix

Template figure B Treatment measurements over time by subject figure

Figure 14.2.4 Urge to use (VAS Score) mean graphs (Full analysis set)

See appendix Template figure C Measurements over time by treatment with confidence interval bars figure

Figure 14.4.1 Individual plasma concentrations over time (lin-log) (Pharmacokinetic analysis set)

See appendix Template figure A Subject measurements over time by treatment figure

Figure 14.4.2 Individual plasma concentrations over time (lin-lin) (Pharmacokinetic analysis set)

See appendix Template figure A Subject measurements over time by treatment figure


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021 45 (49)


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Figure 14.4.3 Mean plasma concentrations over time (lin-log) (Pharmacokinetic analysis set)

See appendix

Template figure B Treatment measurements over time by subject figure

Figure 14.4.4 Mean plasma concentrations over time (lin-lin) (Pharmacokinetic analysis set)

See appendix

Template figure B Treatment measurements over time by subject figure


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

### 14.5 Listings

Listing 16.2.1.1. Discontinued subjects (All subjects)

Listing 16.2.2.1. Protocol deviations (All subjects)

Listing 16.2.3.1 Subjects excluded from PKAS (All subjects)

Listing 16.2.3.2 Population definitions (All subjects)

Listing 16.2.3.3. Non-eligible subjects (All subjects)

Listing 16.2.4.1. Demography (Full analysis set)

Listing 16.2.4.2 Medical/surgical history (Full analysis set)

Listing 16.2.5.1. Prior and concomitant medications (Full analysis set)

Listing 16.2.6.1. Nicotine-use habits (Full analysis set)

Listing 16.2.7.1. HIV, hepatitis B and C (All subjects)

Listing 16.2.8.1. Other laboratory measurements (All subjects)

Listing 16.2.9.2. Product evaluation scale (PES) (Full analysis set)


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Listing 16.2.9.3. Urge to use questionnaire (Full analysis set)

Listing 16.2.9.4. Products preference scale (PPS) (Full analysis set)

Listing 16.2.10.1. Plasma concentration (Pharmacokinetic analysis set)

Listing 16.2.10.2. PK parameters (Pharmacokinetic analysis set)

Listing 16.2.19.1. Nicotine pouch collection (Pharmacokinetic analysis set)

Listing 16.2.12.1. Adverse events, part 1 (Full analysis set)

Listing 16.2.12.2. Adverse events, part 2 (Full analysis set)

Listing 16.2.12.3. Serious adverse events, part 1 (Full analysis set)

Listing 16.2.12.3. Serious adverse events, part 2 (Full analysis set)

Listing 16.2.12.4. Serious adverse events, seriousness criteria (Full analysis set)

Listing 16.2.13.1. Safety laboratory (Full analysis set)

Listing 16.2.14.1. Vital signs (Full analysis set)

Listing 16.2.15.1. ECG (Full analysis set)


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021


Study Code: IB-OND-ZONEX-11 CTC Project No: 369-62-2021

Listing 16.2.16.1. Physical examinations (Full analysis set)

Listing 16.2.17.1. Disposition (All subjects)

Listing 16.2.18.1. Subject visits (All subjects)

Listing 16.2.19.1. Subject elements (All subjects)


Document name: IB-OND-ZONEX-11\_SAP\_v1.0\_10NOV2021